CLINICAL TRIAL: NCT01158573
Title: Role of Cysteinyl Leukotrienes in the Pathogenesis of Asthma in Obesity
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Michael Coffey, Associate Professor Internal Medicine, Pulmonary Division, University of Michigan
Other Study IDs: 36879
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2017-06

CONDITIONS: Asthma; Obesity
Keywords: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Subjects will provide 30 cc of blood, a urine sample and we will collect 1-2 ml. of exhaled breath condensate for analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Healthy non-asthmatic obese adults: Healthy non-asthmatic obese adults
- Healthy non-asthmatic non-obese adults: Healthy non-asthmatic non-obese adults
- Asthmatic obese adults: Asthmatic obese adults
- Asthmatic non-obese adults: Asthmatic non-obese adults

SUMMARY:
The purpose of this study is to examine whether there are higher levels of cysteinyl leukotrienes in obese subjects than in non-obese subjects. Cysteinyl leukotrienes are pro-inflammatory substances that cause asthma by narrowing the airways of the lung. The investigators want to see if subjects with increased fat stores and therefore increased leptin, which is a fat-related protein that regulates leukotrienes, have increased levels of leukotrienes in the blood, lung and urine. The investigators would also like to determine the relationship between cysteinyl leukotrienes and exhaled nitric oxide levels in asthmatics with and without obesity. Nitric oxide is anti-inflammatory and suppresses leukotriene synthesis.

DETAILED DESCRIPTION:
This is a cross-sectional observational study to characterize the association between obese asthmatics and the inflammatory mediators cysteinyl leukotrienes. Our hypothesis is that altered adipokine levels in obesity result in augmented cysteinyl leukotriene synthesis that play a significant role in the pathogenesis of asthma in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yr old adults with asthma, non-smoking for at least one year
* Healthy non-smoking adults, aged 18-65 without asthma
* Heavy subjects with BMI > 30 kg/m2
* Subjects with normal weight (BMI between 20-25 kg/m2)
* Subject not taking anti-leukotriene therapy (Singulair, Accolate, Zyflo)

Exclusion Criteria:

* No chronic oral steroid use
* No recent history of infection
* No recent history of flare of lung disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UM Housing Residents/Student Dorms UM Human Research Recruiting Registry (e.g., ENGAGE - http://www.med.umich.edu/engage/) Department or unit-specific research recruiting registry (provide UM IRB project number below) Other UM subject pools (describe below) Patients or their medical records from the UM Health System or any other UM health care provider (e.g., School of Dentistry, University Health Service, University Center for Language and Literacy)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Coffey, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: OA Obese Asthma BMI >30
  NANO Non asthma non obese
  ANO Asthma non obese
  NAO Non asthma obese BMI >30
  Started July 2010 completed May 2013
Pre-assignment Details: Pre-assignment weight determined and pulmonary function testing prior to enrollment in observational study
  One time point study when mediators were mesaured.
Groups:
- Obese Asthma: Obese Asthma (OA)
  BMI > 30 Obese
  Asthma based on asthma questionnaire, peak flow meter, spirometry, history, physical examination and medication use.
- Non Asthma, Non-obese; Asthma, Non-obese: BMI 20-25 Non obese
- Non Asthma, Obese: BMI .30
Period: Overall Study
Arm/Group | Obese Asthma | Non Asthma, Non-obese | Asthma, Non-obese | Non Asthma, Obese
Started | 30 (Aimed to recruit 160 from July 2010 to May 2013. Each subject studied on one time point only) | 30 | 29 | 28
Completed | 30 (Study completed at 117 subjects.) | 30 | 29 | 28
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Obese Asthma (OA): BMI > 30 Obese
  Asthma based on asthma questionnaire, peak flow meter, spirometry, history, physical examination and medication use.
- Non Asthma Non-obese (NANO): BMI 20-25 Non obese
- Asthma Non Obese (ANO): BMI 20-25 Non obese
  Asthma based on asthma questionnaire, peak flow meter, spirometry, history, physical examination and medication use.
- Non Asthma Obese (NAO): BMI > 30 Obese
- Total: Total of all reporting groups
Arm/Group | Obese Asthma (OA) | Non Asthma Non-obese (NANO) | Asthma Non Obese (ANO) | Non Asthma Obese (NAO) | Total
Number analyzed (Participants) | 30 | 30 | 29 | 28 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (10.3) | 31.5 (11.6) | 29.9 (9.8) | 42.7 (13.6) | 37.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 20 | 21 | 77
  Male | 9 | 15 | 9 | 7 | 40
BMI [Mean (Standard Deviation); unit: kg/m^2] | 38.9 (6.1) | 22.9 (1.7) | 22.8 (1.7) | 37.7 (5.4) | 30.8 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Leptin
Description: Measurement of plasma leptin in obese and non obese asthmatics and non-asthmatic subjects from a single blood draw.
Time Frame: Observational: one time point from a blood draw after more than 6 hours fasting
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Obese Asthma (OA) | Non Asthma Non-obese (NANO) | Asthma Non Obese (ANO) | Non Asthma Obese (NAO)
Number analyzed (Participants) | 30 | 30 | 29 | 28
ng/ml | 55.4 (26.9) | 8.9 (8.8) | 24.2 (12.9) | 46.5 (24.2)
Statistical Analysis 1: Comparison: Obese Asthma (OA) vs Non Asthma Non-obese (NANO) vs Asthma Non Obese (ANO) vs Non Asthma Obese (NAO); Test type: Superiority or Other; p < 0.0001, ANOVA — Hypothesis that leptin levels in OA is not different from the other 3 groups

2. Primary Outcome: Exhaled Nitric Oxide (FeNO)
Description: Exhaled breath nitic oxide ppb (averaged values from 2 exhalations per participant)
Time Frame: Observational: Two exhalations within 1 minute
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Obese Asthma (OA) | Non Asthma Non-obese (NANO) | Asthma Non Obese (ANO) | Non Asthma Obese (NAO)
Number analyzed (Participants) | 30 | 30 | 29 | 28
parts per billion (ppb) | 17.8 (9.3) | 20.7 (14.0) | 29.5 (22.4) | 19.9 (10.4)
Statistical Analysis 1: Comparison: Obese Asthma (OA) vs Non Asthma Non-obese (NANO) vs Asthma Non Obese (ANO) vs Non Asthma Obese (NAO); Test type: Superiority or Other; p = 0.002, ANOVA

3. Primary Outcome: Urine Cysteinyl Leukotriene Per Creatinine
Description: Urine inflammatory mediators measured from a single urine sample
Time Frame: sample taken over 5 minutes or less
Measure: Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | Obese Asthma (OA) | Non Asthma Non-obese (NANO) | Asthma Non Obese (ANO) | Non Asthma Obese (NAO)
Number analyzed (Participants) | 30 | 30 | 29 | 28
pg/mg creatinine | 7.21 (3.2) | 6.35 (3.3) | 6.31 (2.65) | 6.67 (3.3)
Statistical Analysis 1: Comparison: Obese Asthma (OA) vs Non Asthma Non-obese (NANO) vs Asthma Non Obese (ANO) vs Non Asthma Obese (NAO); Test type: Superiority or Other; p = 0.725, ANOVA

4. Primary Outcome: Ratio U Cys-LT/FeNO
Description: Responsiveness to leukotriene modifier medication by measuring the urine cysteinyl leukotriene/exhaled nitric oxide ratio
Time Frame: sample taken over 5 minutes or less
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Obese Asthma (OA) | Non Asthma Non-obese (NANO) | Asthma Non Obese (ANO) | Non Asthma Obese (NAO)
Number analyzed (Participants) | 30 | 30 | 29 | 28
ratio | 0.5 (0.4) | 0.42 (0.3) | 0.3 (0.21) | 0.44 (0.21)
Statistical Analysis 1: Comparison: Obese Asthma (OA) vs Non Asthma Non-obese (NANO) vs Asthma Non Obese (ANO) vs Non Asthma Obese (NAO); Test type: Superiority or Other; p = 0.16, ANOVA

ADVERSE EVENTS:
Arm/Group | Obese Asthma (OA) | Non Asthma Non-obese (NANO) | Asthma Non Obese (ANO) | Non Asthma Obese (NAO)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes